CLINICAL TRIAL: NCT04168333
Title: A Phase I, Single Center, Randomized, Double-blind, Placebo Controlled, Single Dose (SD) and Multiple Dose (MD), Dose-escalation Clinical Trial to Evaluate the Tolerability and Preliminary Antiviral Activity of Therapeutic Hepatitis B Adenovirus Injection (T101) in Chronic Hepatitis B Patients
Brief Title: Safety and Efficacy of Therapeutic Hepatitis B Adenovirus Injection (T101) in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Tianjin Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-2017-001
Record Dates: First submitted 2019-10-24; First posted 2019-11-19 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B Virus (HBV)
Keywords: Hepatitis B virus (HBV) infection
MeSH Terms: conditions — Hepatitis B; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T101 Group (Active Comparator): The study will consist of 2 cohorts:
  Single Dose (SD) Cohort:
  9 chronic hepatitis B patients will be enrolled and be divided into 3 groups, with 3 patients in each group.
  Multiple Dose (MD) Cohort:
  18 chronic hepatitis B patients will be enrolled and be divided into 2 groups, with 9 patients in each group.
  Interventions: Biological: T101 Group
- Placebo Group (Placebo Comparator): The study will consist of 2 cohorts:
  Single Dose (SD) Cohort:
  3 chronic hepatitis B patients will be enrolled in this group.
  Multiple Dose (MD) Cohort:
  6 chronic hepatitis B patients will be enrolled in this group.
  Interventions: Biological: Placebo Group

INTERVENTIONS:
Biological: T101 Group — Single Dose (SD) Cohort:
  In each group, 3 of chronic hepatitis B patients will be subcutaneously injected with different dose level of T101 at 1.0E+9VP (Group1)/1.0E+10VP (Group2)/1.0E+11VP (Group 3) on D1.
  Multiple Dose (MD) Cohort:
  In each group, 9 of chronic hepatitis B patients will be subcutaneously injected with different dose level of T101 at 1.0E+10VP (Group1)/1.0E+11VP (Group2) on D1, D8, D15.
  Arms: T101 Group
Biological: Placebo Group — Single Dose (SD) Cohort:
  3 of chronic hepatitis B patients will be subcutaneously injected with placebo on D1.
  Multiple Dose (MD) Cohort:
  6 of chronic hepatitis B patients will be subcutaneously injected with placebo on D1, D8, D15.
  Arms: Placebo Group

SUMMARY:
Hepatitis B virus (HBV) infection is a worldwide health problem. It has been proved that the persistence of HBV is associated with the failure to stimulate an efficient HBV-specific immune response. T101, the Chinese counterpart of TG1050, is a replication-defective adenovirus serotype 5 (Ad5) expressing multiple HBV-specific antigens (core, polymerase and envelope) and is used as therapeutic vaccine for chronic hepatitis B patients. The application of T101 aims at inducing a broad HBV-specific cellular immune response and ultimately eliminating HBV infection.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, single dose (SD) and multiple dose (MD) administration study.

Primary Objective: Safety and tolerability;

Secondary Objective:

1. Antiviral activity of T101 (HBsAg levels).
2. Cellular (HBV-specific) and humoral (AD5 neutralizing antibodies, NAd5) immune responses to T101.

Key Inclusion Criteria:

1. Chronic hepatitis B patients with positive HBsAg.
2. Patients must be receiving antiviral treatment with nucleoside analogs and have negative HBV DNA (defined as HBV DNA <20 IU/mL).

ELIGIBILITY:
Inclusion Criteria:

* 1) Signed, written Independent Ethics Committee (IEC)-approved informed consent.
* 2) Patients can cooperate to finish the trial in accordance with the requirements of protocol.
* 3）Patients (including partners) are willing to have no pregnancy program and take effective contraceptive measures voluntarily from the initiation of trial to 6 months after the last administration.
* 4) 18 through 65 years of age, inclusive.
* 5）Body weight is no less than 50 kg for male or no less than 45 kg for female and body mass index(BMI) must be within the range of 18-30kg/m2.
* 6）Compensated liver disease; defined as total bilirubin ≤2 × ULN, PT ≤ 1.2 ×ULN, platelets ≥100,000/mm3(100*109/L), serum albumin ≥35 g/L, and no prior history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, variceal hemorrhage).
* 7) Patients must be receiving antiviral treatment with nucleoside analog and have negative HBV DNA(defined HBV DNA <20 IU/Ml).
* 8) Chronic hepatitis B patients have positive HBsAg.
* 9) ALT ≤ 1.5×ULN.
* 10) Haemoglobin ≥ 10 g/L
* 11) Creatinine clearance > 50mL/min.
* 12) Neutrophils ≥1,200/mm3(1.2*109/L).
* 13) FibroScan score ≤ 17.5 kPa within 6 months prior to screening or during screening, or proven not to have cirrhosis according to liver tissues within 12 months.

Exclusion Criteria:

* 1) Addicted to smoking (>5 cigarettes per day) for 3 months prior to the initiation of trial.
* 2) Subjects susceptible to allergies, including a history of allergy to investigational medical product (IMP) or its buffer.
* 3) History of drug abuse and/or alcohol abuse(≥14 units of alcohol per week; 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine).
* 4) Patients who have donated or lost an amount of blood> 450ml within 3 months prior to the screening of the trial.
* 5) Patients who are positive urine test of drug on screening or a history of drug abuse or use of narcotic drugs during the past five years.
* 6) Patients who have used any drug that can alter the enzyme activity of liver within 28 days prior to screening.
* 7) Patients who have taken any prescription, nonprescription, vitamin product or herbal medicine within 14 days prior to the screening(except for nucleoside analogues).
* 8) Patients who have taken a special diet (including dragon fruit, mango, grapefruit, etc.) within 2 weeks prior to screening, or have strenuous exercise, or other factors that affect drug absorption, distribution, metabolism and excretion.
* 9) Patients who are taking inhibitors or inducers of CYP3A4, P-gp or Bcrp such as itraconazole, ketoconazole or dronedarone.
* 10) Patients who have significant changes in diet or exercise habit.
* 11) Patients who have participated in any clinical trial or taken any IMP within 3 months prior to the trial.
* 12) Patients with an clinically significant and abnormal ECG.
* 13) Female patients who are pregnant, breast-feeding or positive result of pregnancy test.
* 14) Patients with abnormal laboratory test results that have clinically significant or clinically significant disease(including but not limited to the gastrointestinal tract, kidney, liver, neurological, haematological, endocrine, lung, immune, mental or cardiovascular disease).
* 15) Patients with α-fetoprotein > 50 ng/Ml.
* 16) Patients with positive hepatitis C antibody, HIV antibody, or Treponema pallidum antibody on screening.
* 17) Patients who could not be enrolled in the judgement of the investigators.
* 18) Patients with acute disease or accompanied medication on screening.
* 19) Patients who have taken chocolate or any food and drink that are rich in caffeine or xanthine within 48 hours prior to the administration of IMP.
* 20) Patients who have taken any alcohol product within 24 hours prior to the administration of IMP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Adverse events | through study completion, an average of 1 year
  Observe all the adverse events of all patients, record their clinical features, severity, time of occurence, end time, duration, treatment measures, recovery and determine their correlation with T101
Vital signs index | Single Dose Group: baseline, Day-1, Day1, Day8, Day15, Day2ine9; Multiple Dose Group: baseline, Day-1, Day7, Day8, Day14, Day15, Day22, Day29, Day43, Day71, Day99.
  vital signs measure: include body temperature, pulse rate, respiratory rate and blood pressure, to observe whether there are abnormal index, especially whether there are abnormal index caused by acute allergic reaction.
Routine blood test | Single Dose Group: baseline, Day-1, Day8, Day15, Day29; Multiple Dose Group: baseline, Day-1, Day7, Day14, Day22, Day29, Day43, Day71, Day99, Day 197, Day379.
  Observe the blood routine tests results of all patients, compare the change of each index before and after the treatment, and determine their correlation with T101 if abnormal index occur.
Blood biochemical test | Single Dose Group: baseline, Day-1, Day8, Day15, Day29; Multiple Dose Group: baseline, Day-1, Day7, Day14, Day22, Day29, Day43, Day71, Day99, Day 197, Day379.
  Observe the blood biochemical tests results of all patients, compare the change of each index before and after the treatment, and determine their correlation with T101 if abnormal index occur.
Coagulation function test | Single Dose Group: baseline, Day-1, Day8, Day15, Day29; Multiple Dose Group: baseline, Day-1, Day7, Day14, Day22, Day29, Day43, Day71, Day99, Day 197, Day379.
  Observe the coagulation function tests results of all patients, compare the change of each index before and after the treatment, and determine their correlation with T101 if abnormal index occur.
Routine urinalysis | Single Dose Group: baseline, Day-1, Day8, Day15, Day29; Multiple Dose Group: baseline, Day-1, Day7, Day14, Day22, Day29, Day43, Day71, Day99, Day 197, Day379.
  Observe the routine urinalysis tests results of all patients, compare the change of each index before and after the treatment, and determine their correlation with T101 if abnormal index occur.

SECONDARY OUTCOMES:
HBsAg quantitative levels | Single Dose Group: Day1, Day29; Multiple Dose Group: Day1, Day29, Day43, Day71, Day99, Day197, Day379.
  Evaluate the efficacy of T101
HBeAg quantitative levels | Single Dose Group: Day1, Day29; Multiple Dose Group: Day1, Day29, Day43, Day71, Day99, Day197, Day379.
  Evaluate the efficacy of T101
Ad5 neutralizing antibodies | Single Dose Group: Day1, Day15, Day29; Multiple Dose Group: Day1, Day29, Day43, Day71, Day99, Day197, Day379.
  Use Analysis of luciferase Ad5 neutralizing antibody method to evaluate the changes of NAd5 titers after T101 administration
Cellular and humoral immune responses | Single Dose Group: Day1, Day15, Day29; Multiple Dose Group: Day1, Day29, Day43, Day71, Day99, Day197, Day379.
  Detect the T-cell responses by interferon-γ（INF-γ） ELISPOT

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, China